CLINICAL TRIAL: NCT01712685
Title: PET Imaging Of Renal Cell Carcinoma With 18F-VM4-037: A Phase II Pilot Study For Detection Of Disease And Correlation With VHL Mutation Status
Brief Title: Imaging Studies of Kidney Cancer Using 18F-VM4-037
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed to accrual because imaging agent was no longer available.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Metwalli, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 130018; 13-C-0018
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoma, Renal Cell; Kidney Neoplasms
Keywords: Kidney Neoplasm; RCC; Biodistribution of 18F-VM4-037; CAIX Staining; Tumor Angiogenesis
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — 3-(4-(2-fluoroethoxy)phenyl)-2-(3-methyl-2-(4-((2-sulfamoylbenzo(d)thiazol-6-yloxy)methyl)-1H-1,2,3-triazol-1-yl)butanamido)propanoic acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Cell Carcinoma (Experimental)
  Interventions: Drug: 18F-VM4-037; Procedure: PET/CT

INTERVENTIONS:
Drug: 18F-VM4-037 — Drug being tested for use in cancer imaging studies. It may help tumor tissue show up more clearly during scans.
Procedure: PET/CT
  Other Names: Positron emission tomography; Computed tomography

SUMMARY:
Background:

- The drug 18F-VM4-037 is being tested for use in cancer imaging studies. It may help tumor tissue show up more clearly during scans. Researchers want to see how well it works for scans for people who have kidney cancer.

Objectives:

- To test the safety and effectiveness of 18F-VM4-037 during imaging studies of kidney cancer.

Eligibility:

- Adults at least 18 years of age with kidney cancer that will be treated with surgery.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have two positron emission tomography (PET) scans of their kidneys. They will have the scans before and after receiving an injection of 18F-VM4-037. The scans will take about 2 hours to complete.
* About 3 weeks after the PET scans, participants will provide tumor tissue samples from their kidneys.
* This is a scanning study only. Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
BACKGROUND:

* Carbonic Anhydrase IX (CA IX) is a hypoxia-inducible enzyme regulated by the Von Hippel Lindau (VHL) protein that is commonly overexpressed in certain malignancies including renal cell carcinoma (RCC) and may have prognostic significance.
* The VHL gene is commonly mutated or inactivated in RCC tumors and VHL activity regulated the expression and activity of not only CAIX but also CAXII as well as other genes critical for tumor angiogenesis such as vascular endothelial growth factor (VEGF), glucose transporter 1 (GLUT1), glucose transporter 3 (GLUT 3) and platelet derived growth factor (PDGF).
* 18F-VM4-037 is an imaging drug product formulation which binds to the active site ligand of CA-IX and also binds to CAXII. We propose to evaluate 18F-VM4-037 as a positron emission imaging (PET) radiopharmaceutical for the in vivo detection of CA-IX and CAXII in renal tumors.

STUDY OBJECTIVES

PRIMARY OBJECTIVE:

* To evaluate the biodistribution of 18F-VM4-037 within tumor and non-tumor tissues.
* To assess safety of 18F-VM4-037 in patients with primary or metastatic RCC.

ELIGIBILITY:

* Subject is greater than or equal to 18 years old, Eastern Cooperative Oncology Group (ECOG) 0-2.
* Subject must have confirmed primary RCC (greater than or equal to 2.5cm) in diameter on conventional imaging modality or extrarenal/extrahepatic RCC lesion (greater than or equal to 1cm).

DESIGN:

- Twenty subjects with primary RCC greater than or equal to 2.5cm in diameter or extrarenal/extrahepatic lesion suspicious for metastatic RCC (greater than or equal to 1cm in diameter) scheduled for clinically indicated surgery or biopsy will undergo dynamic 18F-VM4-037 PET/CT imaging. Results will be compared with pathology.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject is greater than or equal to18 years old.
* Subject must be scheduled to undergo surgery or biopsy for primary renal cell carcinoma (RCC) greater than or equal to 2.5cm in diameter or extrarenal/extrahepatic metastatic RCC lesion (greater than or equal to1cm in diameter) at the National Institutes of Health (NIH) Clinical Center based on imaging within 3 weeks.
* Chemistry parameters: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2 times of the upper limits of normal; total bilirubin, of < 2 times the upper limits of normal or < 3.0 mg/dl in patients with Gilberts syndrome.
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
* Ability to provide informed consent. All subjects must sign an informed consent form indicating their understanding of the investigational nature and risks of the study before any protocol-related studies are performed.
* The subject has a clinically acceptable medical history, physical examination and vital signs findings during the screening period (from within 21 days before administration of 18F-VM4-037). Components of an acceptable medical history include no active infection at the time of enrollment or within 7 days of enrollment, no prior therapy that results in immunocompromise or impaired renal function (serum creatinine within 2 weeks prior to positron emission tomography (PET) imaging less than or equal to1.8 mg/dl and epidermal growth factor receptor (eGFR) must be > 30 ml/min/1.73m^2) or findings indicating an inability to tolerate the requirements for the scan. Previous exposure to immunocompromising therapy does not exclude the patient; patients must have an absolute neutrophil count > 1.5/microL within 2 weeks of PET imaging.
* If female, must have a negative serum human chorionic gonadotropin (HCG) within 24 hours prior to 18F-VM4-037 injection OR be post menopausal for > 2 years OR be surgically sterile.

EXCLUSION CRITERIA:

* Subjects for whom participating would significantly delay the scheduled standard of care therapy.
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics.
* Other medical conditions deemed by the principle investigator (or associates) or sponsor to make the subject ineligible for protocol procedures.
* Female subject is pregnant or nursing
* The site of the target lesion must not have been part of a radiation portal within 6 months of enrollment.
* Subjects having received another investigational agent within 1 month before administration of 18F-VM4-037.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam R Metwalli, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Background] Latif F, Tory K, Gnarra J, Yao M, Duh FM, Orcutt ML, Stackhouse T, Kuzmin I, Modi W, Geil L, et al. Identification of the von Hippel-Lindau disease tumor suppressor gene. Science. 1993 May 28;260(5112):1317-20. doi: 10.1126/science.8493574.
- [Background] Seizinger BR, Rouleau GA, Ozelius LJ, Lane AH, Farmer GE, Lamiell JM, Haines J, Yuen JW, Collins D, Majoor-Krakauer D, et al. Von Hippel-Lindau disease maps to the region of chromosome 3 associated with renal cell carcinoma. Nature. 1988 Mar 17;332(6161):268-9. doi: 10.1038/332268a0. PMID 2894613
- [Result] Turkbey B, Lindenberg ML, Adler S, Kurdziel KA, McKinney YL, Weaver J, Vocke CD, Anver M, Bratslavsky G, Eclarinal P, Kwarteng G, Lin FI, Yaqub-Ogun N, Merino MJ, Linehan WM, Choyke PL, Metwalli AR. PET/CT imaging of renal cell carcinoma with (18)F-VM4-037: a phase II pilot study. Abdom Radiol (NY). 2016 Jan;41(1):109-18. doi: 10.1007/s00261-015-0599-1. PMID 26830617
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0018.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Cell Carcinoma: This is a single arm, phase II trial of a novel radiotracer that is being evaluated for use in patients with kidney cancer. This study is designed to evaluate the imaging characteristics of this drug for detecting specific types of kidney cancer. This is a single administration trial of a single dose of the drug (18F-VM4-037: Drug being tested for use in cancer imaging studies; it may help tumor tissue show up more clearly during scans.) followed by imaging to assess distribution of the drug in normal and tumor tissue.
Period: Overall Study
Arm/Group | Renal Cell Carcinoma
Started | 12
Completed | 11
Not Completed | 1
Not completed — pt declined to participate before trmt | 1

BASELINE CHARACTERISTICS:
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.62 (14.26)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Known Hereditary Renal Cell Carcinoma Mutation [Count of Participants; unit: Participants] — Demographics information of all the accrued 12 patients; one patient did not receive 18F-VM4-037 injection and positron emission tomography (PET) computed tomography (CT) imaging.
  Participants
    Yes (Von Hippel-Lindau) | 5
    No | 7
Clinical Stage [Count of Participants; unit: Participants] — The T category describes the original tumor. T0: No evidence of primary tumor; T1-T4: Size and/or extent of the primary tumor, with higher numbers indicating larger size/extent. The N category describes whether or not the cancer has reached nearby lymph nodes. N0: No regional lymph node involvement (no cancer found in the lymph nodes). The M category tells whether there are distant metastases (spread of cancer to other parts of the body). M0: No distant metastasis (cancer has not spread to other parts of the body); M1: Distant metastasis (cancer has spread to distant parts of the body).
  Participants
    TONOMO | 1
    T1aNOMO | 7
    T3aNOM1 | 2
    T2NOMO1 | 1
    T1bNOMO | 1
Histology [Count of Participants; unit: Participants]
  Renalcyst | 1
  Clear Renal Cell Carcinoma (ccRCC) | 9
  ccRCC with sarcomatoid differentiation | 1
  ccRCC with sarcomatoid features | 1
Grade [Count of Participants; unit: Participants] — The grades range from 0-4 with higher grades indicating greater size and extent of the tumor.
  Participants
    Not Applicable (N/A) | 1
    2 | 8
    3 | 1
    4 | 2
Tumor Size (cm) [Count of Participants; unit: Participants]
  2.0 | 1
  2.7 | 1
  3.3 | 1
  3.4 | 2
  3.5 | 1
  3.6 | 1
  3.7 | 1
  4.0 | 1
  5.8 | 1
  6.89 | 1
  9.3 | 1

OUTCOME MEASURES:

1. Primary Outcome: Level of Uptake of 18F-VM4-037 in Tumor and Non Tumor Tissues, Calculated as Standardized Uptake Values (SUVs)
Description: The primary outcome measure will be assessed from quantitative measurements (e.g., correlate immunohistochemistry (IHC) results with standardized uptake values (SUVs) from positron emission tomography (PET) images) of the level of uptake of tumor and non tumor tissues into each target lesion, calculated as standardized uptake values. Normal renal parenchyma and muscle are both "non-tumor" tissue.
Time Frame: 58 days
Measure: Mean (Standard Error); unit: Standardized uptake value
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
Standardized uptake value
  Tumor tissue | 6.2 (0.25)
  Nontumor tissue | 5.6 (0.20)
  Muscle tissue | 0.6 (0.21)
  Normal kidney tissue | 35 (3.69)

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 58 days
Measure: Number; unit: participants
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
participants | 2

3. Secondary Outcome: Mean Standard Uptake Value (SUV) for All Target Lesions
Description: Mean SUV for all target lesions was assessed by lesion based analysis to obtain SUV mean (the average SUV value within the lesion contour).
Time Frame: Dynamic imaging was performed for the first 45 minutes post injection and whole body imaging was obtained at 60 minutes post injection. Tumors were surgically excised or biopsied within 4 weeks of imaging.
Measure: Mean (Full Range); unit: Standard uptake value (SUV)
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
Standard uptake value (SUV) | 3.04 [0.58 to 9.61]

4. Secondary Outcome: Mean Standard Uptake Value (SUV) for Primary Clear Cell Renal Carcinoma (ccRCC)
Description: Mean SUV for primary clear cell renal carcinoma was assessed by lesion based analysis to obtain SUV mean (the average SUV value within the lesion contour).
Time Frame: as for outcome 3
Population: Mean SUV for ccRCC after excluding Bosnial 3 Cyst (e.g. Bosnial 3 complex cyst) in one participant.
Measure: Mean (Full Range); unit: Standard uptake value (SUV
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
Standard uptake value (SUV | 2.55 [0.58 to 4.23]

5. Secondary Outcome: Mean Standard Uptake Value (SUV) for Normal Kidney
Description: Mean SUV for normal kidney was assessed by lesion based analysis to obtain SUV mean (the average SUV value within the lesion contour).
Time Frame: as for outcome 3
Measure: Mean (Full Range); unit: Standard uptake value (SUV
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
Standard uptake value (SUV | 35.4 [19.6 to 50.3]

6. Secondary Outcome: Number of Participants With a Mutation of the Von Hippel-Lindau (VHL) Gene
Description: Germline VHL mutation testing was performed using Clinical Laboratory Improvement Amendments (CLIA) certified laboratories.
Time Frame: 21 days prior to enrollment until closure of the study, approximately 14 months.
Population: 5/11 participants had germline VHL testing with 4 having identifiable mutations of the VHL gene. 6/11 participants did not have germline VHL mutation testing due to low index of clinical suspicion although 2/6 had germline analysis for other gene mutations linked to familial renal cell carcinoma conditions.
Measure: Number; unit: participants
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
participants | 4

7. Secondary Outcome: Distribution Volume Ratio (DVR) for the Primary Kidney Lesions
Description: DVR of the lesions was measured by the Logan graphical analysis method.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Distribution volume ratio
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
Distribution volume ratio | 5.2 (2.8)

8. Secondary Outcome: Time to Peak Activity Derived From Time Activity Curve (TAC)
Description: The time to peak activity of radiotracer (tumor marker) uptake indicates the optimal time to image to obtain best tumor visibility.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
Minutes | 9.08 (3.06)

9. Secondary Outcome: Kinetic (Ki) Rate Constant
Description: Ki was assessed by the Patlak graphical analysis method which measures the uptake rate constant Ki.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1/Minutes
Arm/Group | Renal Cell Carcinoma
Number analyzed (Participants) | 11
1/Minutes
  Primary kidney lesions | 0.01 (.05)
  Normal kidney | .45 (0.22)
  Liver | 0.54 (0.18)

ADVERSE EVENTS:
Arm/Group | Renal Cell Carcinoma
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Cell Carcinoma (N=11)
Dysgeusia (Nervous system disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed to accrual because imaging agent was no longer available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No